CLINICAL TRIAL: NCT04248608
Title: Perioperative Analgesic Modalities for Breast Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, lecturer of anesthesia and pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP1907-50101
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Morphine; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- erector spinae block (Experimental): Ultrasound guided erector spinae block with will be done after induction of intravenous anesthesia. After identification of trapezius, rhomboid major, and erector spinae muscles. The needle will be inserted in a cephalad-to-caudal direction until the tip contact transverse process and the needle tip is visualized in the plane deep to the erector spinae muscle. The needle tip position is confirmed by visualizing linear spread of test dose between the muscles after injection. A total dose of 25 mL of 0.25% bupivacaine will be injected.
  Interventions: Procedure: erector spinae block
- serratus anterior block (Experimental): Ultrasound guided serratus anterior block will be done after induction of intravenous anesthesia. The serratus anterior, latissimus dorsi, and the intercostal muscles will be identified in the fourth and fifth intercostal level, an 18 G Tuohy needle will be advanced in the plane between the serratus anterior muscle and the intercostal muscles. A total dose of bupivacaine 25ml in a concentration of 0.25% will be administered under the serratus muscle after a test dose using an in-plane technique.
  Interventions: Procedure: serratus plane block
- intravenous morphine (Active Comparator): intravenous morphine will be administrated in a dose of 0.1 mg per kg after induction of general anesthesia
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Procedure: serratus plane block — ultrasound guided block
  Other Names: SAPB
  Arms: serratus anterior block
Procedure: erector spinae block — ultrasound guided block
  Other Names: ESPB
  Arms: erector spinae block
Drug: Morphine Sulfate — intravenous morphine sulfate 0.1 mg/kg
  Other Names: opioid
  Arms: intravenous morphine

SUMMARY:
The incidence of breast cancer is among women world wide, detection increased with introduction of mammography as a screening tool. surgical resection of breast cancer contributes to the generation of acute and chronic post mastectomy pain. This study aims at comparing the effect of erector spinae block versus serratus block versus intravenous morphine in patients undergoing modified radical mastectomy for breast cancer surgeries regarding pain control and possible side effects

DETAILED DESCRIPTION:
One of the most common types of cancer affecting women is breast cancer. Surgical resection is one of the main approaches applied for solid tumors. surgical approach for breast cancer involve the breast region. Various analgesic modalities are used for proper perioperative pain control. Morphine has always been considered as the gold standard analgesic, however opioids have multiple side effects. Several loco-regional techniques have been introduced for breast surgery pain management including serratus plane block (SPB) and erector spinae plane (ESP) block. In this study the investigators are comparing the effect of erector spinae block versus serratus block versus intravenous morphine in patients undergoing modified radical mastectomy for breast cancer surgeries regarding intraoperative and postoperative analgesia, time to first analgesic, any possible side effects

ELIGIBILITY:
Inclusion Criteria:

* female 18-65 years old patients undergoing modified radical mastectomy

Exclusion Criteria:

* patient refusal, local infection at site of block coagulation defect abnormal kidney or liver functions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | 24 hours
  minimum score (0), maximum score (10) maximum score (10)
Total morphine consumption | 24 hours
  total morphine in mg received in first 24 hours postoprative
First time to receive morphine | 24 hours
  first time to receive morphine in the postoperative period (first 24 hours)

SECONDARY OUTCOMES:
mean arterial blood pressure | 24 hours
  hemodynamic parameters
heart rate | 24 hours
  hemodynamic parameters

CONTACTS AND LOCATIONS:
Overall Officials: walaa Y Elsabeeny, MD, Principal Investigator — Lecturer
Locations (1):
- Department of anesthesia and pain medicine. National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elsabeeny WY, Shehab NN, Wadod MA, Elkady MA. Perioperative Analgesic Modalities for Breast Cancer Surgeries: A Prospective Randomized Controlled Trial. J Pain Res. 2020 Nov 12;13:2885-2894. doi: 10.2147/JPR.S274808. eCollection 2020. PMID 33209056